CLINICAL TRIAL: NCT07072585
Title: A Phase 2/3 Randomized Trial Investigating Daratumumab on a Modified Augmented BFM (aBFM) Backbone in Newly Diagnosed T-Lymphoblastic Leukemia (T-ALL) and T-Lymphoblastic Lymphoma (T-LL)
Brief Title: Testing the Addition of Daratumumab to Chemotherapy for Treating Patients With Newly-Diagnosed T-Cell Lymphoblastic Leukemia (T-ALL) and T-Cell Lymphoblastic Lymphoma (T-LL)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL2331; NCI-2025-02230 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL2331 (Other: Children's Oncology Group); AALL2331 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2025-05-07; First posted 2025-07-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Stage II T Lymphoblastic Leukemia/Lymphoma; Stage III T Lymphoblastic Leukemia/Lymphoma; Stage IV T Lymphoblastic Leukemia/Lymphoma; T Acute Lymphoblastic Leukemia; T Lymphoblastic Lymphoma
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Biopsy; Specimen Handling; Bortezomib; calaspargase pegol; Asparaginase; Cyclophosphamide; Cytarabine; daratumumab; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Spinal Puncture; Magnetic Resonance Spectroscopy; Mercaptopurine; Methotrexate; merphos; Methylprednisolone; exifone; Medrol Veriderm; nelarabine; pegaspargase; Prednisolone; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Hydrocortisone; Thioguanine; High-Energy Shock Waves; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group I, Arm A (T-ALL, no daratumumab) (Active Comparator): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Nelarabine; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate
- Group I, Arm B (T-ALL, daratumumab) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Biological: Daratumumab; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Nelarabine; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate
- Group II, Arm C (T-LL, no daratumumab) (Active Comparator): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Drug: Bortezomib; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate
- Group II, Arm D (T-LL, daratumumab) (Experimental): See Detailed Description
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Bone Scan; Drug: Bortezomib; Drug: Calaspargase Pegol; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Cytarabine; Biological: Daratumumab; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Mercaptopurine Oral Suspension; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Pegaspargase; Procedure: Positron Emission Tomography; Drug: Prednisolone; Drug: Prednisone; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Procedure: Ultrasound Imaging; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
  Arms: Group II, Arm C (T-LL, no daratumumab); Group II, Arm D (T-LL, daratumumab)
Drug: Bortezomib — Given IV or SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
  Arms: Group II, Arm C (T-LL, no daratumumab); Group II, Arm D (T-LL, daratumumab)
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: Group II, Arm C (T-LL, no daratumumab); Group II, Arm D (T-LL, daratumumab)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IT or IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Daratumumab — Given IV
  Other Names: Daratumumab Biosimilar HLX15; Daratumumab-fihj; Darzalex; HLX15; HuMax-CD38; JNJ 54767414; JNJ-54767414; JNJ54767414
  Arms: Group I, Arm B (T-ALL, daratumumab); Group II, Arm D (T-LL, daratumumab)
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Lumbar Puncture — Under lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mercaptopurine Oral Suspension — Given PO
  Other Names: 6-MP Oral Suspension; Purixan; Xaluprine
Drug: Methotrexate — Given IT or IV or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Drug: Nelarabine — Given IV
  Other Names: 2-Amino-6-methoxypurine arabinoside; 506U78; Arranon; Compound 506U78; GW506U78
  Arms: Group I, Arm A (T-ALL, no daratumumab); Group I, Arm B (T-ALL, daratumumab)
Drug: Pegaspargase — Given IV or IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Procedure: Positron Emission Tomography — Undergo PET or PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: Group II, Arm C (T-LL, no daratumumab); Group II, Arm D (T-LL, daratumumab)
Drug: Prednisolone — Given PO or IV
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
Drug: Prednisone — Given PO or IV
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II/III trial tests the addition of daratumumab to chemotherapy for treating patients with newly-diagnosed T-ALL and T-LL. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Chemotherapy drugs work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with daratumumab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the event-free survival (EFS) from the end of induction (EOI) in patients with newly diagnosed T-ALL who are randomized to either receive a modified augmented Berlin-Frankfurt-Münster (aBFM) chemotherapy backbone or a modified aBFM backbone with the addition of daratumumab.

II. To compare the EFS from the EOI in patients with newly diagnosed T-LL who are randomized to a modified aBFM chemotherapy backbone with bortezomib or to a modified aBFM backbone with bortezomib and the addition of daratumumab.

SECONDARY OBJECTIVES:

I. To compare health-related quality of life (HRQoL) and therapy-related toxicity and tolerability between patients with T-ALL or T-LL randomized to a modified aBFM backbone or to a modified aBFM backbone with the addition of daratumumab.

II. To compare overall survival (OS) from date of randomization in patients with newly diagnosed T-ALL who are randomized to either receive a modified aBFM chemotherapy backbone or a modified aBFM backbone with the addition of daratumumab.

III. To compare OS from date of randomization in patients with newly diagnosed T-LL who are randomized to a modified aBFM chemotherapy backbone with bortezomib or to a modified aBFM backbone with bortezomib and the addition of daratumumab.

EXPLORATORY OBJECTIVES:

I. In patients with newly diagnosed T-LL, to determine if minimal residual disease (MRD) testing at EOI can predict EFS and/or OS.

II. In T-ALL patients, to describe changes in the immunophenotype (specifically CD38 surface expression on T-ALL/T-LL blasts) and for the development of anti-daratumumab antibodies over the course of treatment and correlate changes with clinical outcomes and demographic variables.

III. To explore the associations between family-reported social determinants of health and both clinical outcomes (including incidence of treatment-related toxicities, EFS, OS), and leukemia/lymphoma and host biology.

IV. To describe outcome differences (EFS and OS) in patients with T-LL who differ in degrees of positron emission tomography (PET)-imaging avid disease at the EOI.

V. To explore potential imaging findings and biomarkers of significant/severe nelarabine-induced central nervous system toxicities by central review of magnetic resonance imaging (MRI) and to investigate possible clinical features in patients experiencing such toxicities.

VI. To bank peripheral blood specimens for future correlative studies in patients with T-LL.

VII. To compare EFS and OS from the EOI in patients with newly diagnosed T-ALL who are MRD positive (≥ 0.01%) at the EOI to those who are MRD negative at the EOI.

OUTLINE: This is a phase II study, followed by a phase III study. Patients are assigned to 1 of 2 groups.

GROUP I T-ALL:

INDUCTION: Patients receive cytarabine intrathecally (IT) once at the time of lumbar puncture, or day 1, daunorubicin intravenously (IV) over 1 - 15 minutes on days 1, 8, 15 and 22, dexamethasone orally (PO) or IV twice a day (BID) on days 1 - 28, vincristine IV on days 1, 8, 15 and 22, pegaspargase IV over 1 - 2 hours or intramuscularly (IM) once on day 4 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 4, and methotrexate IT on days 8 and 29 (patients with central nervous system [CNS]1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 8, 15, 22 and 29 (patients with CNS3). Induction treatment continues over 35 days in the absence of disease progression or unacceptable toxicity.

EOI: Patients are randomized to 1 of 2 arms.

ARM A:

CONSOLIDATION: Patients receive nelarabine IV over 60 minutes QD on days 1 - 5 and 36 - 40, cyclophosphamide IV over 30 - 60 minutes on days 8 and 43, cytarabine IV over 1 - 30 minutes or subcutaneously (SC) QD on days 8 - 11, 15 - 18, 43 - 46 and 50 - 53, mercaptopurine PO QD on days 8 - 21 and 43 - 56, methotrexate IT on days 15, 22, 50 and 57 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 15, 22, 50 and 57 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM on days 22 and 57 or calaspargase pegol-mknl IV over 1 - 2 hours on days 22 and 57, and vincristine IV on days 22, 29, 57 and 64. Patients with persistent testicular disease undergo radiation therapy QD for 12 fractions within the first two weeks of consolidation. Consolidation treatment continues over 77 days in the absence of disease progression or unacceptable toxicity. Patients with MRD < 1% following consolidation proceed to interim maintenance.

INTERIM MAINTENANCE: Patients receive methotrexate IT on days 1 and 31 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 1 and 31 (patients with CNS3), methotrexate IV over 2 - 15 minutes on days 1, 11, 21, 31 and 41, pegaspargase IV over 1 - 2 hours or IM on days 2 and 22 or calaspargase pegol-mknl IV over 1 - 2 hours on days 2 and 23, and vincristine IV on days 1, 11, 21, 31 and 41. Interim maintenance treatment continues over 56 days in the absence of disease progression or unacceptable toxicity. Patients with MRD < 0.1% following interim maintenance proceed to delayed intensification.

DELAYED INTENSIFICATION:

PART 1: Patients receive dexamethasone PO or IV BID on days 1 - 7 and 15 - 21, doxorubicin IV over 3 - 15 minutes on days 1, 8 and 15, methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM once on day 4 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 4, and vincristine IV on days 1, 8 and 15. Delayed intensification part 1 treatment continues over 28 days in the absence of disease progression or unacceptable toxicity.

PART 2: Patients receive nelarabine IV over 60 minutes QD on days 29 - 33, cyclophosphamide IV over 30 - 60 minutes once on day 36, cytarabine IV over 1 - 30 minutes or SC QD on days 36 - 39 and 43 - 46, thioguanine PO QD on days 36 - 49, methotrexate IT on days 36 and 43 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 36 and 43 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM once on day 50 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 50, and vincristine IV on days 50 and 57. Delayed intensification part 2 treatment continues over 35 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE:

CYCLES 1 - 3: Patients receive methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), mercaptopurine PO QD on days 1 - 28 and 36 - 84, prednisone PO or IV BID on days 1 - 5 and 57 - 61 or prednisolone PO or IV BID on days 1 - 5 and 57 - 61 or methylprednisolone IV BID on days 1 - 5 and 57 - 61, vincristine IV on days 1 and 57, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71 and 78, and nelarabine IV over 60 minutes QD on days 29 - 33. Cycles repeat every 84 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 4 +: Patients receive methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), prednisone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61 or prednisolone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61, mercaptopurine PO QD on days 1 - 84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71 and 78. Cycles repeat every 84 days until 2 years from the start of interim maintenance in the absence of disease progression or unacceptable toxicity.

ARM B:

CONSOLIDATION: Patients receive daratumumab IV on days 8, 15, 22, 29, 43, 50, 57 and 64, nelarabine IV over 60 minutes QD on days 1 - 5 and 36 - 41, cyclophosphamide IV over 30 - 60 minutes on days 8 and 43, cytarabine IV over 1 - 30 minutes or SC QD on days 8 - 11, 15 - 18, 43 - 46 and 50 - 53, mercaptopurine PO QD on days 8 - 21 and 43 - 56, methotrexate IT on days 15, 22, 50 and 57 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 15, 22, 50 and 57 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM on days 23 and 58 or calaspargase pegol-mknl IV over 1 - 2 hours on days 23 and 58, and vincristine IV on days 22, 29, 57 and 64. Patients with persistent testicular disease undergo radiation therapy QD for 12 fractions within the first two weeks of consolidation. Consolidation treatment continues over 77 days in the absence of disease progression or unacceptable toxicity. Patients with MRD < 1% following consolidation proceed to interim maintenance.

INTERIM MAINTENANCE: Patients receive daratumumab IV on days 1, 21 and 41, methotrexate IT on days 1 and 31 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 1 and 31 (patients with CNS3), methotrexate IV over 2 - 15 minutes on days 1, 11, 21, 31 and 41, pegaspargase IV over 1 - 2 hours or IM on days 2 and 22 or calaspargase pegol-mknl IV over 1 - 2 hours on days 2 and 23, and vincristine IV on days 1, 11, 21, 31 and 41. Interim maintenance treatment continues over 56 days in the absence of disease progression or unacceptable toxicity. Patients with MRD < 0.1% following interim maintenance proceed to delayed intensification.

DELAYED INTENSIFICATION:

PART 1: Patients receive daratumumab IV on days 1 and 15, dexamethasone PO or IV BID on days 1 - 7 and 15 - 21, doxorubicin IV over 3 - 15 minutes on days 1, 8 and 15, methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), vincristine IV on days 1, 8 and 15, and pegaspargase IV over 1 - 2 hours or IM once on day 4 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 4. Delayed intensification part 1 treatment continues over 28 days in the absence of disease progression or unacceptable toxicity.

PART 2: Patients receive nelarabine IV over 60 minutes QD on days 29 - 33, daratumumab IV on days 36 and 50, cyclophosphamide IV over 30 - 60 minutes once on day 36, cytarabine IV over 1 - 30 minutes or SC QD on days 36 - 39 and 43 - 46, thioguanine PO QD on days 36 - 49, methotrexate IT on days 36 and 43 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 36 and 43 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM once on day 51 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 51, and vincristine IV on days 50 and 57. Delayed intensification part 2 treatment continues over 35 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE:

CYCLES 1 - 3: Patients receive methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), mercaptopurine PO QD on days 1 - 28 and 36 - 84, prednisone PO or IV BID on days 1 - 5 and 57 - 61 or prednisolone PO or IV BID on days 1 - 5 and 57 - 61 or methylprednisolone IV BID on days 1 - 5 and 57 - 61, vincristine IV on days 1 and 57, methotrexate PO on days 8, 15, 22, 36, 43, 50, 57, 64, 71 and 78, and nelarabine IV over 60 minutes QD on days 29 - 33. Cycles repeat every 84 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

CYCLES 4 +: Patients receive methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), prednisone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61 or prednisolone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61, mercaptopurine PO QD on days 1 - 84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71 and 78. Cycles repeat every 84 days until 2 years from the start of interim maintenance in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo echocardiography (ECHO) during screening and bone marrow biopsy and aspiration as well as lumbar puncture throughout the study. Patients may undergo MRI, ultrasound and biopsy on study as well as may undergo blood sample collection throughout the study.

GROUP II T-LL:

INDUCTION: Patients receive bortezomib IV over 3 - 5 seconds or SC on days 1, 4, 8 and 11, cytarabine IT once at the time of lumbar puncture, or day 1, daunorubicin IV over 1 - 15 minutes on days 1, 8, 15 and 22, prednisone PO or IV BID on days 1 - 28 or prednisolone PO or IV BID on days 1 - 28 or methylprednisolone IV BID on days 1 - 28, methotrexate IT on days 8 and 29 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 8, 15, 22 and 29 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM once on day 4 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 4, and vincristine IV on days 1, 8, 15 and 22. Induction treatment continues over 35 days in the absence of disease progression or unacceptable toxicity.

EOI: Patients are randomized to 1 of 2 arms.

ARM C:

CONSOLIDATION: Patients receive cyclophosphamide IV over 30 - 60 minutes on days 1 and 29, cytarabine IV over 1 - 30 minutes or SC QD on days 1 - 4, 8 - 11, 29 - 32 and 36 - 39, mercaptopurine PO QD on days 1 - 14 and 29 - 42, methotrexate IT on days 1, 8, 15 and 22 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 1, 8, 15 and 22 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM on days 15 and 43 or calaspargase pegol-mknl IV over 1 - 2 hours on days 15 and 43, and vincristine IV on days 15, 22, 43 and 50. Patients with persistent testicular disease undergo radiation therapy QD for 12 fractions within the first two weeks of consolidation. Consolidation treatment continues over 63 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) following consolidation proceed to interim maintenance.

INTERIM MAINTENANCE: Patients receive methotrexate IT on days 1 and 31 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 1 and 31 (patients with CNS3), methotrexate IV over 2 - 15 minutes on days 1, 11, 21, 31 and 41, pegaspargase IV over 1 - 2 hours or IM on days 2 and 22 or calaspargase pegol-mknl IV over 1 - 2 hours on days 2 and 23, and vincristine IV on days 1, 11, 21, 31 and 41. Interim maintenance treatment continues over 56 days in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION:

PART 1: Patients receive bortezomib IV over 3 - 5 seconds or SC on days 1, 4, 15 and 18, dexamethasone PO or IV BID on days 1 - 7 and 15 - 21, doxorubicin IV over 3 - 15 minutes on days 1, 8 and 15, methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), vincristine IV on days 1, 8 and 15, and pegaspargase IV over 1 - 2 hours or IM once on day 4 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 4. Delayed intensification part 1 treatment continues over 28 days in the absence of disease progression or unacceptable toxicity.

PART 2: Patients receive cyclophosphamide IV over 30 - 60 minutes once on day 29, cytarabine IV over 1 - 30 minutes or SC QD on days 29 - 32 and 36 - 39, thioguanine PO QD on days 29 - 42, methotrexate IT on days 29 and 36 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 29 and 36 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM once on day 43 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 43, and vincristine IV on days 43 and 50. Delayed intensification part 2 treatment continues over 28 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), mercaptopurine PO QD on days 1 - 84, prednisone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61 or prednisolone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61 or methylprednisolone IV BID on days 1 - 5, 29 - 33 and 57 - 61, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71 and 78. Cycles repeat every 84 days for 2 years from the start of interim maintenance in the absence of disease progression or unacceptable toxicity.

ARM D:

CONSOLIDATION: Patients receive daratumumab IV on days 1, 8, 15, 22, 29, 36, 43 and 50, cyclophosphamide IV over 30 - 60 minutes on days 1 and 29, cytarabine IV over 1 - 30 minutes or SC QD on days 1 - 4, 8 - 11, 29 - 32 and 36 - 39, mercaptopurine PO QD on days 1 - 14 and 29 - 42, methotrexate IT on days 1, 8, 15 and 22 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 1, 8, 15 and 22 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM on days 16 and 44 or calaspargase pegol-mknl IV over 1 - 2 hours on days 16 and 44, and vincristine IV on days 15, 22, 43 and 50. Patients with persistent testicular disease undergo radiation therapy QD for 12 fractions within the first two weeks of consolidation. Consolidation treatment continues over 63 days in the absence of disease progression or unacceptable toxicity. Patients with a CR following consolidation proceed to interim maintenance.

INTERIM MAINTENANCE: Patients receive daratumumab IV on days 1, 21 and 41, methotrexate IT on days 1 and 31 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT on days 1 and 31 (patients with CNS3), methotrexate IV over 2 - 15 minutes on days 1, 11, 21, 31 and 41, pegaspargase IV over 1 - 2 hours or IM on days 2 and 22 or calaspargase pegol-mknl IV over 1 - 2 hours on days 2 and 23, and vincristine IV on days 1, 11, 21, 31 and 41. Interim maintenance treatment continues over 56 days in the absence of disease progression or unacceptable toxicity.

DELAYED INTENSIFICATION:

PART 1: Patients receive daratumumab IV on days 1 and 15, bortezomib IV over 3 - 5 seconds or SC on days 1, 4, 15 and 18, dexamethasone PO or IV BID on days 1 - 7 and 15 - 21, doxorubicin IV over 3 - 15 minutes on days 1, 8 and 15, methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), vincristine IV on days 1, 8 and 15, and pegaspargase IV over 1 - 2 hours or IM once on day 4 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 4. Delayed intensification part 1 treatment continues over 28 days in the absence of disease progression or unacceptable toxicity.

PART 2: Patients receive daratumumab IV QD on days 29 and 43, cyclophosphamide IV over 30 - 60 minutes once on day 29, cytarabine IV over 1 - 30 minutes or SC QD on days 29 - 32 and 36 - 39, thioguanine PO QD on days 29 - 42, methotrexate IT QD on days 29 and 36 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT QD on days 29 and 36 (patients with CNS3), pegaspargase IV over 1 - 2 hours or IM once on day 44 or calaspargase pegol-mknl IV over 1 - 2 hours once on day 44, and vincristine IV QD on days 43 and 50. Delayed intensification part 2 treatment continues over 28 days in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive methotrexate IT once on day 1 (patients with CNS1 or CNS2) or methotrexate IT, hydrocortisone IT and cytarabine IT once on day 1 (patients with CNS3), mercaptopurine PO QD on days 1 - 84, prednisone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61 or prednisolone PO or IV BID on days 1 - 5, 29 - 33 and 57 - 61 or methylprednisolone IV BID on days 1 - 5, 29 - 33 and 57 - 61, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71 and 78. Cycles repeat every 84 days for 2 years from the start of interim maintenance in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo ECHO during screening and lumbar puncture as well as computed tomography (CT) or MRI, PET or PET-CT or bone scan throughout the study. Patients may undergo ultrasound and biopsy on study as well as may undergo blood sample collection and bone marrow biopsy and aspiration throughout the study.

After completion of study treatment, patients are followed up for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be enrolled on APEC14B1 and consented to eligibility screening (part A) prior to treatment and enrolled on AALL2331.
* Patients must be > 365 days and < 21 years of age at the time of diagnosis.
* * Newly diagnosed T-cell acute lymphoblastic leukemia (T-ALL) or T-lineage lymphoblastic lymphoma (T-LL) stages II-IV.

  * Note: A diagnosis of T-ALL is established when leukemic blasts lack myeloperoxidase or evidence of B-lineage derivation (CD19/CD22/CD20), and express either surface or cytoplasmic CD3 or two or more of the antigens CD8, CD7, CD5, CD4, CD2 or CD1a, and are present either in peripheral blood or > 25% in the bone marrow. If surface CD3 is expressed on all leukemic cells, additional markers of immaturity, including TdT, CD34 or CD99 will be assessed for expression. Cases with uncertain expression will receive additional review within the appropriate Children's Oncology Group (COG) reference laboratory.
  * For T-LL patients with tissue available for flow cytometry, the criterion for diagnosis should be analogous to T-ALL. For tissue processed by other means (i.e. paraffin blocks), the methodology and criteria for immunophenotypic analysis to establish the diagnosis of T-LL defined by the submitting institution will be accepted.

Exclusion Criteria:

* Diagnosis of Down syndrome (trisomy 21).
* Patients with known Charcot-Marie-Tooth disease.
* * Patients must not have received any cytotoxic chemotherapy for either the current diagnosis of T-ALL, T-LL or for any cancer diagnosis prior to the initiation of protocol therapy on AALL2331 with the exception of:

  * Steroid pretreatment: Prednisone or methylprednisolone for ≤ 120 hours (5 days) in the 7 days prior to initiating induction chemotherapy or for ≤ 336 hours (14 days) in the 28 days prior to initiation of protocol therapy does not affect eligibility.
  * Intrathecal cytarabine; or
  * Pretreatment with hydroxyurea; or
  * 600 cGy of chest irradiation, if medically necessary.
  * Pre-treatment with dexamethasone in the 28 days prior to initiation of protocol therapy is not allowed with the exception of a single dose of dexamethasone used during sedation to prevent or treat airway edema. Patients who receive a single dose of dexamethasone to prevent or treat airway edema in the 28 days preceding diagnosis are eligible for this study.
* * Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.

  * Lactating females who plan to breastfeed their infants.
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation.
* Known severe persistent asthma anytime in the previous two years or uncontrolled asthma of any classification.
* Peripheral neurotoxicity: Pre-existing ≥ grade 2 sensory or motor peripheral neurotoxicity.
* Seizure disorder: Patients must not have an uncontrolled seizure disorder. Patients with a seizure history or a controlled seizure disorder are eligible. A controlled seizure disorder is defined as having stable or decreasing symptoms over the past 3 months without anti-epileptic medications or is on a stable or decreasing dose of anti-epileptic medication.
* * Patients who are previously known to be seropositive for HIV except for HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of enrollment on this trial.

  * Patients with evidence of chronic hepatitis B (HBV) infection, except for patients who have an HBV viral load that is undetectable on suppressive therapy.
  * Patients with a history of hepatitis C virus (HCV) infection, except for those patients who have been treated and cured, or patients who are currently on HCV treatment who have an undetectable HCV viral load.
* Patients with significant hepatic dysfunction defined as those with an alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) > 10x upper limit of normal (ULN) or direct bilirubin > 2x ULN unless the patient has known Gilbert's syndrome or has hepatic involvement from leukemic or lymphomatous infiltration.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Ages: 365 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1708 (Estimated)
Dates: Start 2026-06-28 (Estimated); Primary Completion 2035-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) in patients with newly diagnosed T-cell lymphoblastic leukemia (T-ALL) | From date of randomization (randomization conducted at the end of induction [EOI]) to date of first event (consolidation failure, interim maintenance failure, relapse, secondary malignant neoplasm [SMN], death from any cause), assessed up to 4 years
  Will compare EFS in patients with newly diagnosed T-ALL who are randomized to either receive a modified augmented Berlin-Frankfurt-Munich (aBFM) chemotherapy backbone or a modified aBFM backbone with the addition of daratumumab. Patients without an EFS event will be censored at the date of last follow-up. The survival time analyses assume a Weibull distribution with a shape parameter of 0.45 (based on historical controls). A phase 2/3 design will be used.
EFS in patients with newly diagnosed T-cell lymphoblastic lymphoma (T-LL) | From date of randomization (randomization conducted at the EOI) to date of first event (consolidation failure, relapse, progressive disease, SMN, death from any cause), assessed up to 4 years
  Will compare EFS in patients with newly diagnosed T-LL who are randomized to a modified aBFM chemotherapy backbone with bortezomib or to a modified aBFM backbone with bortezomib and the addition of daratumumab. Patients without an EFS event will be censored at the date of last follow-up. The survival time analyses assume a Weibull distribution with a shape parameter of 0.45 (based on historical controls).

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) | Baseline (at time of randomization) to day 64 of consolidation
  Will compare HRQoL between patients with T-ALL or T-LL randomized to a modified aBFM backbone or to a modified aBFM backbone with the addition of daratumumab. Will use the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Global Health scale (PGH-7). The PROMIS PGH-7 has a standard deviation of 10 points, with higher scores indicating better HRQoL.
Incidence of therapy-related toxicity and tolerability | Assessed up to 3 cycles post randomization (each cycle is approximately 2-3 months)
  Will compare therapy-related toxicity and tolerability between patients with T-ALL or T-LL randomized to a modified aBFM backbone or to a modified aBFM backbone with the addition of daratumumab. Will be assessed for all patients and the rates compared between the randomized arms (T-ALL: arm A versus (vs) arm B and T-LL: arm C vs arm D). Rates by arm will be reviewed by the study committee on a monthly basis and will also be provided in the biannual reports to the Children's Oncology Group Data and Safety Monitoring Committee for review. Any concerns regarding excessive rates of any toxicities will be discussed in the context of any required therapy modifications.
Overall survival (OS) in patients with newly diagnosed T-ALL | From date of randomization (randomization conducted at the EOI) to date of death (death due to any cause), assessed up to 4 years
  Will compare OS in patients with newly diagnosed T-ALL who are randomized to either receive a modified aBFM chemotherapy backbone or a modified aBFM backbone with the addition of daratumumab. Patients who are alive will be censored at date of last follow-up. Comparison of OS between the two randomized arms will be conducted at the time of the final analysis for the primary objective (EFS). Analyses will be based on stratified log-rank tests. In addition, descriptive OS rates post randomization will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto. In particular, 4-year OS rates in arm A and arm B will be estimated. Estimation of treatment effect will be done using intent-to-treat (ITT) analysis. Hazard ratio (HR) and the confidence interval will be estimated based on Cox regression models as appropriate.
Overall survival (OS) in patients with newly diagnosed T-LL | From date of randomization (randomization conducted at the EOI) to date of death (death due to any cause), assessed up to 4 years
  Will compare OS in patients with newly diagnosed T-LL who are randomized to a modified aBFM chemotherapy backbone with bortezomib or to a modified aBFM backbone with bortezomib and the addition of daratumumab. Patients who are alive will be censored at date of last follow-up. Comparison of OS between the two randomized arms will be conducted at the time of the final analysis for the primary objective (EFS). Analyses will be based on log-rank tests. In addition, descriptive OS rates post randomization will be estimated using the Kaplan-Meier method and standard errors and confidence intervals estimated by the method of Peto. In particular, 4-year OS rates in arm C and arm D will be estimated. Estimation of treatment effect will be done using ITT analysis. HR and the confidence interval will be estimated based on Cox regression models as appropriate.

OTHER OUTCOMES:
EFS from end of induction patients with newly diagnosed T-LL | Assessed up to 4 years
  Will determine if minumal residual disease (MRD) testing in patients with newly diagnosed T-LL at EOI can predict EFS. EFS will be compared for T-LL patients with negative MRD (defined as < 0.1%) and those who with MRD ≥ 0.1% at the EOI. EFS will be defined as time from the EOI to date of first event (consolidation failure, relapse, progressive disease, SMN, death from any cause), and patients without an EFS event will be censored at the date of last follow-up. In addition, comparison of EFS by the EOI MRD status (positive vs negative) will be conducted among randomized patients. Comparisons will be conducted by treatment arms. A potential interaction between MRD at the EOI with treatment arms will be assessed.
OS from end of Induction in patients with newly diagnosed T-LL | Assessed up to 4 years
  Will determine if MRD testing in patients with newly diagnosed T-LL at EOI can predict OS. OS will be compared for T-LL patients with negative MRD (defined as < 0.1%) and those who with MRD ≥ 0.1% at the EOI. OS will be defined as time from the EOI to date of death, with patients who are alive being censored at date of last follow-up. In addition, comparison of OS by the EOI MRD status (positive vs negative) will be conducted among randomized patients. Comparisons will be conducted by treatment arms. A potential interaction between MRD at the EOI with treatment arms will be assessed.
Immunophenotype in T-ALL patients | Assessed at baseline, end of Induction (Induction is 29 days), and relapse (up to 10 years)
  Will describe changes in T-ALL patients in the immunophenotype (specifically CD38 surface expression on T-ALL/T-LL blasts) correlate changes with clinical outcomes and demographic variables. Differences between patients treated with daratumumab and those who are not treated with daratumumab will be assessed; the comparisons between arm A and arm B will be based on test of proportions, Fisher's exact test or logistic regression, as appropriate.
Development of anti-daratumumab antibodies in T-ALL patients | Assessed up to 3 years
  Will describe the development of anti-daratumumab antibodies over the course of treatment and correlate changes with clinical outcomes and demographic variables. Analyses will be restricted to T-ALL patients randomized to arm B. Analyses will be based on test of proportions, Fisher exact test, logistic regression, log-rank test, semi-parametric or parametric survival analysis, as appropriate.
Family-reported social determinants of health | Up to approximately 1 year of treatment
  Will describe family-reported social determinants of health and assess its association with clinical outcomes (including incidence of treatment-related toxicities, EFS, OS), and leukemia/lymphoma and host biology. These analyses will be based on analysis of variance, test of proportions, logistic regression, log-rank test, semi-parametric or parametric survival analysis methods, etc., as appropriate.
EFS from date of PET scan at the end of induction in patients with T-LL | Assessed up to 4 years
  Will describe outcome differences (EFS) in patients with T-LL who differ in degrees of positron emission tomography (PET)-imaging avid disease at the EOI. EFS will be compared for T-LL patients with a positive PET scan (Deauville 4 and 5) to patients with a negative PET scan (Deauville 1, 2 and 3) at the EOI. EFS will be defined as time from date of PET scan (i.e., EOI) to date of first event (relapse, consolidation failure, progressive disease, SMN, death from any cause); patients without an EFS event will be censored at the date of last follow-up. EFS will be presented based on Kaplan-Meier method. Comparisons of EFS between PET positive and PET negative groups will be performed using log-rank test, semi-parametric or parametric survival analysis methods, as appropriate.
OS from date of PET scan at the end of Induction in patients with newly diagnosed T-LL | Assessed up to 4 years
  Will describe outcome differences (OS) in patients with T-LL who differ in degrees of PET-imaging avid disease at the EOI. OS will be compared for T-LL patients with a positive PET scan (Deauville 4 and 5) to patients with a negative PET scan (Deauville 1, 2 and 3) at the EOI. OS will be defined as time from date of PET scan to date of death, with patients who are alive censored at the date of last follow-up. OS curves will be presented based on Kaplan-Meier method. Comparisons of EFS/OS between PET positive and PET negative groups will be performed using log-rank test, semi-parametric or parametric survival analysis methods, as appropriate.
Magnetic resonance imaging (MRI) imaging findings associated with onset of seizure or grade 3 or higher neurotoxicity attributed to treatment with nelarabine | Assessed to the end of protocol therapy, up to 3 years.
  Will explore potential MRI imaging findings that are associated with severe nelarabine-induced central nervous system toxicities. In T-ALL patients that experience any new onset seizure or grade 3 or higher neurotoxicity attributed to treatment with nelarabine, results of MRI imaging and other biomarkers associated with toxicity and associations with clinical features will be described to determine potential risk factors. These analyses will be based on analysis of variance, test of proportions, log-rank test, semi-parametric or parametric survival analysis methods, etc., as appropriate. MRI findings will be analyzed to identify a pathognomonic signal of nelarabine neurotoxicity. In addition it is anticipated that MRIs obtained for this purpose will have signals which will exclude neurotoxic events related to non-nelarabine therapeutics.
Peripheral blood specimens in patients with T-LL | Up to 10 years
  Will bank peripheral blood specimens for future correlative studies in patients with T-LL.
EFS from end of induction in patients with newly diagnosed T-ALL | Assessed up to 4 years
  Will compare EFS from the EOI in patients with newly diagnosed T-ALL who are MRD positive (≥ 0.01%) at the EOI to those who are MRD negative at the EOI. EFS will be defined as time from the EOI to date of first event (consolidation failure, interim maintenance failure, relapse, SMN, death from any cause), and patients without an EFS event will be censored at the date of last follow-up. In addition, comparison of EFS by the EOI MRD status (positive vs negative) will be conducted among randomized patients (n=874, all of them should have the EOI MRD tested). For this comparison, EFS will be defined as time from date of randomization to date of first event (consolidation failure, interim maintenance failure, relapse, SMN, death from any cause), and patients without an EFS event will be censored at the date of last follow-up.
OS from end of Induction in patients with newly diagnosed T-ALL | Assessed up to 4 years
  Will compare OS from the EOI in patients with newly diagnosed T-ALL who are MRD positive (≥ 0.01%) at the EOI to those who are MRD negative at the EOI. OS will be defined as time from the EOI to date of death, with patients who are alive being censored at date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Keith J August, Principal Investigator — Children's Oncology Group